CLINICAL TRIAL: NCT01440348
Title: Simultaneous Multiple Cruciate Ligament Reconstructions Using a Single Achilles Allograft
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Police Hospital (Other Government)
Responsible Party: Principal Investigator, Jung Ho Noh, Orthopaedic surgeon, National Police Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPH2010-001
Record Dates: First submitted 2011-09-21; First posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Rupture of Posterior Cruciate Ligament; Rupture of Anterior Cruciate Ligament
Keywords: Achilles allograft; cruciate ligament; reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Achilles allograft (Experimental)
  Interventions: Procedure: cruciate ligament reconstruction

INTERVENTIONS:
Procedure: cruciate ligament reconstruction — Multiple cruciate ligament reconstructions with a single Achilles allograft with was divided into two or three strips according to the thickness and length of the allograft.

SUMMARY:
This study introduce cases of simultaneous multiple cruciate ligament reconstructions with a single free tendon Achilles allograft using new technique.

ELIGIBILITY:
Inclusion Criteria:

* subjects who had any concomitant meniscus or cartilage injuries

Exclusion Criteria:

* subjects who required reconstruction of medial or lateral collateral ligament, or posterolateral ligament complex
* subject who wanted reconstruction with autograft
* subject who denied participation in this study
* subject who would meet the national reimbursement criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
circumference and length of the Achilles allograft | day 1
  After the fresh frozen Achilles allograft was thawed, circumference and length of the tendinous portion of the allograft were measured. According to the circumference and length of the allograft, it was divided into two or three grafts for cruciate ligament reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Ho Noh, M.D., Ph.D., Principal Investigator — National Police Hospital
Locations (1):
- National Police Hospital, Seoul, South Korea